CLINICAL TRIAL: NCT04811976
Title: The Effects of Anxiety and Depression on Stent Restenosis in Patients With Acute Coronary Syndrome After Percutaneous Coronary Intervention
Brief Title: The Relationship Between Anxiety, Depression and Stent Restenosis After Percutaneous Coronary Intervention
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021W123
Record Dates: First submitted 2021-03-20; First posted 2021-03-23 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Coronary Heart Disease; Percutaneous Coronary Intervention
Keywords: In-stent restenosis; Coronary heart disease; Anxiety state; Depressive slale
MeSH Terms: conditions — Coronary Disease; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Percutaneous coronary intervention is currently one of the effective methods for the treatment of ACS. Unfortunately, the incidence of ISR is as high as 10%-20% at 3-6 months after PCI. So it is necessary to identify the potential risk factors to provide evidence for the prevention of ISR. Current research shows that anxiety and depression are related to the increased risk of major adverse cardiac events and mortality in patients with acute myocardial infarction. But there remains a relative paucity of evidence for the association between anxiety and depression and in-stent restenosis (ISR) .So a retrospective cohort study was conducted in the first hospital of Qinhuangdao in 2015-2020. The patients who underwent coronary angiography 1 year after PCI in our hospital from January 2015 to September 2020 were selected. Patients were divided into ISR and non-ISR groups depending on the follow-up coronary angiography results. Logistic regression model was utilized for analyzing the association of depression and anxiety with the in-stent restenosis (ISR) after PCI.

DETAILED DESCRIPTION:
Percutaneous coronary intervention is currently one of the effective methods for the treatment of ACS. Unfortunately, postoperative in-stent restenosis (ISR) is still inevitable. The incidence of ISR is as high as 10%-20% at 3-6 months after PCI. And its prevention and treatment is very difficult clinical problems. So it is necessary to identify the potential risk factors to provide evidence for the prevention of ISR. Current research shows that anxiety and depression are related to the increased risk of major adverse cardiac events and mortality in patients with acute myocardial infarction. But there remains a relative paucity of evidence for the association between anxiety and depression and in-stent restenosis (ISR) .

A retrospective cohort study was conducted in the first hospital of Qinhuangdao in 2015-2020. The patients who underwent coronary angiography 1 year after PCI in our hospital from January 2015 to September 2020 were selected. Patients were divided into ISR and non-ISR groups depending on the follow-up coronary angiography results. Every 3 months until 12 months, the patients were consecutively recruited and followed up. Anxiety and depression were assessed using the Zung self-rating anxiety scale (SAS), self-rating depression scale (SDS) and psychosomatic symptom scale at each follow-up timepoint. Relative clinical information was recorded and analyzed. Logistic regression model was utilized for analyzing the association of depression and anxiety with the in-stent restenosis (ISR) after PCI.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of acute coronary syndrome The degree of coronary artery stenosis is greater than 90% The degree of coronary artery stenosis is greater than 75% and there is evidence of ischemia

Exclusion Criteria:

Patients who did not receive stents for the first time Patients who had undergone coronary artery bypass grafting Patients with stent implantation due to stent stenosis Patients who had stents implanted for chronic complete coronary artery occlusion Patients with malignant tumors Patients with autoimmune diseases Patients with severe hepatic and renal insufficiency Patients with cardiomyopathy Patients with congenital heart disease Patients with valvular disease Patients present with acute stress events

Ages: 55 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients who underwent coronary angiography 1 year after PCI in the first hospital of Qinhuangdao from January 2015 to September 2020 were selected. Patients were divided into ISR and non-ISR groups depending on the follow-up coronary angiography results. Every 3 months until 12 months, the patients were consecutively recruited and followed up. Anxiety and depression were assessed using the Zung self-rating anxiety scale (SAS), self-rating depression scale (SDS) and psychosomatic symptom scale at each follow-up timepoint.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
In-stent restenosis | 1 year
  Because of the recurrence of symptoms, patients who have done the PCI more than 12 months do the coronary angiography in our hospital. Two interventionists were assigned to record the coronary angiography and complete the corresponding diagnosis in an independent way. If there was a difference in diagnosis, a third doctor was assigned to perform the correlation analysis and analyze and process the other data of the study subjects by blind method. In-stent restenosis was defined asin-stenosis of lumen diameter ≥50% occurred in the diseased vessels, including the coronary arteries in the stent and at both ends of the stent ≤5 mm from the edge of the stent.

SECONDARY OUTCOMES:
Other adverse cardiac events | 1 year
  Including death, recurrent myocardial infarction, and recurrent angina

CONTACTS AND LOCATIONS:
Locations (1):
- 中国, Qinhuangdao, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided